CLINICAL TRIAL: NCT02927652
Title: Evaluating Psychiatric Comorbidity in Otolaryngology
Brief Title: Psychiatric Comorbidity
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00075353
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Otorhinolaryngologic Diseases
MeSH Terms: conditions — Otorhinolaryngologic Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaires for new patients: New patients seen at Duke Clinic for Head and Neck Surgery & Communication Sciences or Duke Raleigh Otolaryngology will be administered questionnaires (BSI-18, CG-CAHPS, and patient control scale).
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — New patients at the Duke Clinic 1F and Duke Raleigh Otolaryngology will be asked to complete the Brief Symptom Inventory-18 (BSI-18), patient control scale, and CG-CAHPS.
  If a patients answers a 1, 2, 3, or 4 to question #17 ("Thoughts of ending your life") on the BSI-18, the nurse will immediately contact the investigator, who will refer for further assessment and/or treatment. The Duke Social Work office is available to provide support, and the Duke Emergency Department has certified social workers and a psychiatric team to do full evaluations if needed.

SUMMARY:
The goals of this project are aimed at the following:

1. Identifying psychiatric comorbidity in patients presenting to the HNSCS clinic 1F and Duke Otolaryngology of Raleigh clinic using the validated assessment tool Brief Symptom Inventory (BSI-18) and the patient control scale. The BSI-18 is an 18 question and patient control an 8 item tool that takes about four minutes to complete.
2. Gathering data regarding patient satisfaction in new patients to the HNSCS clinics via the CG-CAHPS visit survey.
3. Examining relationships between psychiatric comorbidity and patient satisfaction.
4. Examining relationships between psychiatric comorbidity and healthcare system use.

DETAILED DESCRIPTION:
Patients with multiple otolaryngology complaints experience psychosocial distress. This psychosocial distress can have an adverse effect on treatment outcomes for the primary complaint and on the overall patient experience. It can result in greater costs for more care that may not be best-directed. This has implications not only for the patients, but also for providers' quality metrics.

Data will be collected via surveys and a chart review. New patients at the Duke Clinic 1F and Duke Raleigh Otolaryngology will be asked to complete the BSI-18, patient control scale, and disease specific outcome measure upon patient intake by the clinic nurse. The CG-CAHPS Visit Survey 2.1 will be completed at the conclusion of the clinical encounter. Patient participation consists of these surveys on their initial visit only.

The PI and/or a resident will conduct a chart review of these patients looking for history of psychiatric diagnoses and/or related prescriptions. Patients who have psychiatric diagnoses and/or prescriptions in the chart will be considered to have their needs "met", in that they are receiving care. Data regarding diagnoses and prescriptions will also be entered into REDCap.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* New patient appointment at Duke Clinic 1F or Duke Raleigh Otolaryngology
* Ability to read, write, and understand English

Exclusion Criteria:

* Less than 18 years old
* Unable to read, write, and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New patients being seen at Duke Head and Neck Surgery & Communication Sciences (Clinic 1F) or Duke Raleigh Otolaryngology
Sampling Method: Non-Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Identification of psychiatric comorbidity | day 1
  Measured by the Brief Symptom Inventory (BSI-18) questionnaire using a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely). Maximum global severity index of 72. Higher scores indicate psychosocial distress.
Identification of psychiatric comorbidity | day 1
  Measured by the Perceived Control Scale (PCS) questionnaire using a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree).

SECONDARY OUTCOMES:
Patient satisfaction of provider visitCG-CAHPS score | day 1
  Assessment of patient satisfaction measured by CG-CAHPS visit survey. Will be correlated with BSI-18 during data analysis to evaluate whether evidence of psychosocial distress and perception of satisfaction may be correlated.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Cohen, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center and affiliated practices, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided